CLINICAL TRIAL: NCT02366442
Title: Exploring Relationships Among Balance Performance, Cognitive Dysfunction, Affective Dysregulation, and Community Integration in Veterans With Traumatic Brain Injury (TBI)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Azadeh M. Leland, Fellow at polytrauma/TBI at DCVAMC, Washington D.C. Veterans Affairs Medical Center
Other Study IDs: WashingtonVAMC
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Traumatic Brain Injury; TBI
Keywords: dual/multitasking; Executive function; Affective function; Balance
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Whole-Body Irradiation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Exploring relationships among balance performance, cognitive dysfunction, affective dysregulation, and community integration in Veterans with Traumatic Brain Injury (TBI).

SUMMARY:
The overarching goal of the proposed study, named SYNERGY, is to explore relationships among balance performance, cognitive function, affective dysregulation, as they relate to the community re-integration in Veterans with TBI. The SYNERGY study findings can aid in the development of a better outcome models for the clinicians in facilitating effective community re-integration in Veterans with TBI

DETAILED DESCRIPTION:
Examine if there are associations among balance, cognitive and affective function during multitasking activities in Veterans with the diagnosis of TBI.

To determine if an association exists between balance performance and the degree of community re-integration in Veterans with TBI.

To determine which of the three systems, balance performance, cognitive dysfunction or affective dysregulation, is the strongest predictor of community re-integration in Veterans with TBI.

ELIGIBILITY:
Exclusion-inclusion criteria Inclusion Criteria: Enrolled participants will be Veterans with TBI between18 to55 years of age. We identified a wide age range in order to include Veterans from the Iraq and Afghanistan conflicts, as well as Veterans of the Vietnam War. This feature of the inclusion criteria is important since barriers to community re-integration may be affected by impaired balance, cognitive dysfunction, affective dysregulation, across the age spectrum. Consequently, the study findings will potentially benefit not only young Veterans, but also middle aged Veterans.

The Military Acute Concussion Evaluation (MACE): We will use MACE scores of 21/30 to ensure the participants have the cognitive ability to understand our study protocol, and therefore, participate voluntarily in the study. 62 Exclusion Criteria: We will use an exclusion criteria of 12/24 on the Dynamic gait index (DGI) to ensure that patients are ambulatory either with or without the use of assistive device to be able to measure dynamic balance accurately.16 Past Medical History: The following diagnoses will be cause for exclusion -- peripheral neuropathy, Parkinson syndromes, multiple sclerosis; bipolar, schizophrenia, seizure or psychiatric illnesses.

Medically stable patients: It is essential to minimize future medical adverse conditions and minimize the risk of drop out. Therefore, no patient shall be considered for enrollment if they do not meet inclusion/exclusion criteria or have not been recommended by the polytrauma staff at VA DCMC.

The result of VHA TBI Comprehensive Evaluation electronic template will be reviewed following IRB approved and HIPAA compliant data collection procedures. The TBI diagnosis will be obtained from patient's chart review of problem section and physician's notes.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with the diagnosis of TBI
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Exploring relationships among balance performance, cognitive dysfunction, affective dysregulation, and community integration in Veterans with Traumatic Brain Injury (TBI). | 1-2 year